CLINICAL TRIAL: NCT00000773
Title: Phase I Safety and Pharmacokinetics Study of Microparticulate Atovaquone (m-Atovaquone; 566C80) in HIV-Infected and Perinatally Exposed Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: ACTG 227; 11204 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Antifungal Agents; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Biological Availability; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Atovaquone

INTERVENTIONS:
Drug: Atovaquone

SUMMARY:
To determine the safety, tolerance, and pharmacokinetics of a new improved microparticulate suspension formulation of atovaquone administered at one of two dose levels (per 09/30/94 amendment, a third dose level was added) daily for 12 days in HIV-infected and perinatally exposed (per 8/9/95 amendment) infants and children who are at risk of developing Pneumocystis carinii pneumonia (PCP).

Atovaquone has shown prophylactic potential in adults in the treatment of PCP but is poorly absorbed in tablet form. To improve the bioavailability of atovaquone, a new formulation has been prepared as a microparticulate suspension. Since studies in adults have demonstrated substantial safety of this drug, evaluation in children is being pursued.

DETAILED DESCRIPTION:
Atovaquone has shown prophylactic potential in adults in the treatment of PCP but is poorly absorbed in tablet form. To improve the bioavailability of atovaquone, a new formulation has been prepared as a microparticulate suspension. Since studies in adults have demonstrated substantial safety of this drug, evaluation in children is being pursued.

Three cohorts of four patients each (ages 2-12 years, 3 months to less than 2 years, and 1 month to less than 3 months) receive atovaquone daily for 12 days. The oldest age group is treated first. In the absence of unacceptable toxicity, the dose of atovaquone is escalated in subsequent 4-patient cohorts representing each of the age stratifications and (per 9/30/94 amendment) in a separate 4-patient cohort aged 3 months to less than 2 years. If two of four patients in a given cohort experience unacceptable toxicity at the initial dose, two additional patients in the same age range are entered. Blood samples are drawn for pharmacokinetic evaluation. Patients are followed to day 24. Per 9/30/94 amendment, patients aged 3 months to less than 2 years of age who received one of the lower doses may re-enroll in the higher dose cohort after a 1-month washout.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Dideoxycytidine (zalcitabine; ddC).
* Didanosine (ddI).
* Nonaminoglycoside, nonmacrolide, and nonsulfonamide antibiotics.
* Factor VIII.
* IVIG.

Patients must have:

* AIDS, documented HIV infection, perinatal exposure to HIV, or risk of developing PCP.
* Normal EKG and chest radiograph.
* No blood or protein on urinalysis.
* Consent of parent or guardian.

Prior Medication:

Allowed:

* Prophylactic TMP/SMX if given no less than 3 days prior to study entry.
* Prophylactic aerosolized pentamidine (or a single intravenous dose of 4.0 mg/kg pentamidine) if given no less than 7 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Anticipated organ system or laboratory abnormalities (other than immune system abnormalities) from the primary disease and its treatment during the study.
* Acute or chronic infections requiring treatment during the study. NOTE:
* Thrush and herpes labialis are allowed if these conditions do not require treatment.
* Diarrhea or vomiting.

Concurrent Medication:

Excluded:

* Trimethoprim/sulfamethoxazole.
* Sulfadoxine and pyrimethamine (Fansidar).
* Primaquine.
* Aspirin.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Sulfonamides.
* Dapsone.
* Benzodiazepines.
* Rifampin.
* Erythromycin, clarithromycin, and azithromycin.
* Digitalis.
* Para-aminosalicylic acid (PAS).
* Isoniazid.
* Anticoagulants.
* Any other investigational therapies.

Patients with the following prior condition are excluded:

* History of G6PD deficiency.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hughes W, Study Chair; Dorenbaum A, Study Chair
Locations (6):
- United States (5):
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Dorenbaum A, Sadler BM, Xu J, Van Dyke RB, Wei LJ, Moye J, McNamara J, Yogev R, Diaz C, Hughes W. Phase I safety and pharmacokinetics (PK) study of micronized atovaquone (m-ATQ) in HIV exposed or infected infants and children. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:117 (abstract no 288)